CLINICAL TRIAL: NCT04723420
Title: Pneumatic Retinopexy for Primary Rhegmatogenous Retinal Detachment: To Steamroll or Not
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Kenneth Eng, Pneumatic Retinopexy for Primary Rhegmatogenous Retinal Detachment: To Steamroll or Not, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 270-2019
Record Dates: First submitted 2020-12-19; First posted 2021-01-25 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Rhegmatogenous Retinal Detachment
Keywords: Pneumatic Retinopexy; Steamroll; Direct to break
MeSH Terms: interventions — Fluorescent Antibody Technique, Direct

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Steamroller Technique (Active Comparator): Following intravitreal gas injection, patient positioned face down for 4-6 hours and subsequently patient changes the position of the head so that the bubble is then placed directly over the retina break.
  Interventions: Other: Steamroller technique
- Direct Technique (Active Comparator): Following intravitreal gas injection, patient is immediately positioned so that the bubble is placed directly over the retina break.
  Interventions: Other: Direct technique

INTERVENTIONS:
Other: Steamroller technique — Following intravitreal gas injection, patient positioned face down for 4-6 hours and subsequently patient changes the position of the head so that the bubble is then placed directly over the retina break.
  Arms: Steamroller Technique
Other: Direct technique — Following intravitreal gas injection, patient is immediately positioned so that the bubble is placed directly over the retina break.
  Arms: Direct Technique

SUMMARY:
This is a randomized controlled trial comparing displacement of macula and the rapidity of reattachment of macula between two different positioning techniques after pneumatic retinopexy : Direct technique (patient is positioned so that the bubble is immediately placed directly over the retina break) and Steamroller technique (patient is initially positioned face down for 4-6 hours and subsequently changes their head position so that the bubble is then placed directly over the retina break).

DETAILED DESCRIPTION:
Pneumatic retinopexy (PR) is an established treatment for rhegmatogenous retinal detachment (RRD). In our centre, PR is the most commonly performed procedure for primary RRD repair with a high retinal reattachment success rate. In this procedure, patients are required to position according to the site of pathology following injection of an intravitreal gas bubble. Some practitioners position the patient so that the gas bubble is immediately apposed directly against the retinal break (direct technique). Others favour the steamroller technique whereby the patient is initially positioned face down, then after 4-6 hours, the position is changed sequentially so that the bubble is rolled over the retina towards the break responsible for the detachment (steamroller technique). Variable visual acuity (VA) outcomes and metamorphopsia are common post-procedure complaints despite successful RRD repair with PR. It has been suggested that variability in functional outcomes may be associated with the timing and ease of reattachment of macula. The purpose of this prospective study is to evaluate whether the steamroller technique is superior to the direct technique in faster reattachment of macula with less macula displacement.

ELIGIBILITY:
Inclusion Criteria:

* Primary RRD
* Causative breaks over superior 8 clock hours
* Single break or group of breaks
* No or min proliferative vitreoretinopathy (PVR) (Grade A or B)
* Other breaks or lattice in attached retina are allowed

Exclusion Criteria:

* Retinal break in the inferior 4 clock hours in detached retina
* PVR Grade C or worse
* Significant media opacity (Vitreous hemorrhage, dense cataract, cornea scar, etc)
* Pre-existing ocular pathology [macula hole (MH), epiretinal membrane (ERM), cystoid macula edema (CME), age-related macula degeneration, myopic degeneration, advanced glaucoma, uveitis, amblyopia etc] or previous eye trauma with poor baseline vision
* Previous pars plana vitrectomy
* Age ≤18years old
* Inadequate physical or mental competence to maintain the required postoperative head position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2023-12-07 (Estimated); Study Completion 2023-12-07 (Estimated)

PRIMARY OUTCOMES:
Macular status at Day 1 | 24hours post intervention
  Assessment of macular status by optical coherence tomography at 24 hours after intervention to see which technique is most effective for reattaching the macula

SECONDARY OUTCOMES:
Anatomical displacement of macula and its changes with time. | 1,2, 3 and 6 months post intervention
  Measurement of retinal vessel imprinting on fundus autofluorescence
Functional displacement of macula and its changes with time. | 1,2, 3 and 6 months post intervention
  Measurement of metamorphopsia with M-charts
Macular Status | 1hour, 2hours, Day 2, Week 1, Week 2
  Looking at macula status via optical coherence tomography after intervention to see which technique is more effective in reattaching the macula early
Visual acuity | 1, 3 and 6 months post intervention
  ETDRS
Primary anatomical success | 1, 3 and 6 months post intervention
  Complete reattachment of retina via clinical fundus examination and optos fundus photography

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Eng, MD FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada